CLINICAL TRIAL: NCT00012610
Title: Efficacy of Telepsychiatry in the Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACC 97-034
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Telepsychiatry

INTERVENTIONS:
Procedure: Telepsychiatry

SUMMARY:
Telepsychiatry is a novel means of providing expert psychiatric treatment to patients who live far from a source of care. If it can be demonstrated that treatment via telepsychiatry is as effective as in-person treatment, then many individuals with psychiatric illness will have easy access to psychiatric care, even if they live in geographically remote areas.

DETAILED DESCRIPTION:
Background:

Telepsychiatry is a novel means of providing expert psychiatric treatment to patients who live far from a source of care. If it can be demonstrated that treatment via telepsychiatry is as effective as in-person treatment, then many individuals with psychiatric illness will have easy access to psychiatric care, even if they live in geographically remote areas.

Objectives:

The major goal of this study was to determine whether treatment of depressive disorders via telepsychiatry is as effective as in-person treatment. In addition, this study was designed to determine if depressed patients are as compliant and as satisfied with telepsychiatry as with in-person treatment. Another goal was to compare the cost and cost-effectiveness of remote treatment via telepsychiatry to in-person treatment.

Methods:

In this randomized controlled trial, veterans who presented with depression to any of three VA Maryland Health Care facilities with a SCID-IV depression diagnosis and a Hamilton Rating Scale for Depression (Ham-D) score of 16 or above were eligible for participation. Eligible veterans were randomized to either "in-person" treatment or "remote" treatment. Treatment occurred over six months and consisted of psychotropic medication and psycho-education concerning the disease, medications, and side effects. The major outcome variables included changes in Ham-D depression ratings and Beck Depression Inventory (BDI) self-reported depression ratings.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Depression, Hamilton 16 or above, SCID-IV depression diagnosis

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Ruskin, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States